CLINICAL TRIAL: NCT01813604
Title: Phase III Clinical Trial to Assess the Immunogenicity of a Sequential Dose of Fractional Inactivated Polio Vaccine (f-IPV) and Oral Polio Vaccine (OPV)
Brief Title: Immunogenicity of Inactivated and Live Polio Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Ministry of Health and Family Welfare, Bangladesh (Unknown); NanoPass Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICDDRB-RRC-PR-12028
Record Dates: First submitted 2013-03-12; First posted 2013-03-19 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-03

CONDITIONS: Poliomyelitis
Keywords: Polio; Inactivated polio vaccine; oral polio vaccine; vaccine trial
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group A: Trivalent Oral Polio Vaccine (Active Comparator): Group A will receive 3 doses of trivalent oral polio vaccine (tOPV) at 6, 10 and 14 weeks of age. A challenge dose of tOPV will be administered at 18 weeks of age.
  Interventions: Biological: Group A: Trivalent Oral Polio Vaccine
- Group B: Bivalent Oral Polio Vaccine (Active Comparator): Group B will receive 3 doses of bivalent oral polio vaccine (bOPV) at 6, 10 and 14 weeks of age. A challenge dose of tOPV will be administered at 18 weeks of age.
  Interventions: Biological: Group B: Bivalent Oral Polio Vaccine
- Group C: Inactivated Polio Vaccine (Active Comparator): Group C will receive 2 doses of inactivated polio vaccine (IPV) at 6 and 14 weeks of age. IPV will be administered intramuscularly using standard needle and syringe. A challenge dose of tOPV will be administered at 18 weeks of age.
  Interventions: Biological: Group C: Inactivated Polio Vaccine
- Group D: fractional IPV (f-IPV) (Active Comparator): Group D will receive 2 doses of fractional inactivated polio vaccine (f-IPV) at 6 and 14 weeks of age. f-IPV (one-fifth dose of IPV) will be administered intradermally using MicroJet 600 microneedle hub by NanoPass Technologies. A challenge dose of tOPV will be administered at 18 weeks of age.
  Interventions: Biological: Group D: fractional IPV (f-IPV)
- Arm E: f-IPV and bOPV (Active Comparator): Group E will receive 2 doses of f-IPV at 6 and 14 weeks of age with bOPV at 10 weeks of age. f-IPV will be administered intradermally using MicroJet 600 microneedle hub by NanoPass Technologies. A challenge dose of tOPV will be administered at 18 weeks of age.
  Interventions: Biological: Arm E: f-IPV and bOPV

INTERVENTIONS:
Biological: Group A: Trivalent Oral Polio Vaccine — Group A will receive 3 doses of trivalent oral polio vaccine (tOPV) at 6, 10 and 14 weeks of age. A challenge dose of tOPV will be administered at 18 weeks of age.
  Arms: Group A: Trivalent Oral Polio Vaccine
Biological: Group B: Bivalent Oral Polio Vaccine — Group B will receive 3 doses of bivalent oral polio vaccine (bOPV) at 6, 10 and 14 weeks of age. A challenge dose of tOPV will be administered at 18 weeks of age.
  Arms: Group B: Bivalent Oral Polio Vaccine
Biological: Group C: Inactivated Polio Vaccine — Group C will receive 2 doses of inactivated polio vaccine (IPV) at 6 and 14 weeks of age. IPV will be administered intramuscularly using standard needle and syringe. A challenge dose of tOPV will be administered at 18 weeks of age.
  Arms: Group C: Inactivated Polio Vaccine
Biological: Group D: fractional IPV (f-IPV) — Group D will receive 2 doses of fractional inactivated polio vaccine (f-IPV) at 6 and 14 weeks of age. f-IPV (one-fifth dose of IPV) will be administered intradermally using MicroJet 600 microneedle hub by NanoPass Technologies. A challenge dose of tOPV will be administered at 18 weeks of age.
  Arms: Group D: fractional IPV (f-IPV)
Biological: Arm E: f-IPV and bOPV — Group E will receive 2 doses of f-IPV at 6 and 14 weeks of age with bOPV at 10 weeks of age. f-IPV will be administered intradermally using MicroJet 600 microneedle hub by NanoPass Technologies. A challenge dose of tOPV will be administered at 18 weeks of age.
  Arms: Arm E: f-IPV and bOPV

SUMMARY:
This study is an open-label phase III randomized clinical trial that would compare immunogenicity after receiving one of five different combinations of polio vaccines. Infants will be enrolled and randomized at 6 weeks of age to one of five different arms:

A) Three doses of trivalent oral poliovirus vaccine (tOPV) at 6, 10 and 14 weeks of age B) Three doses of bivalent OPV (bOPV) at 6, 10 and 14 weeks of age C) Two doses of intramuscular (IM) inactivated poliovirus vaccine (IPV) at 6 and 14 weeks of age D) Two doses of intra-dermal (ID) fractional IPV (f-IPV) at 6 and 14 weeks of age E) Sequential administration of ID f-IPV at 6 and 14 weeks of age with bOPV at 10 weeks of age To assess the immunogenicity of each study vaccine and vaccination schedule, antibody titers against poliovirus types 1, 2 and 3 will be determined in sera extracted from blood collected before (at 6 weeks of age) and after receiving 3 doses of study vaccine (18 weeks of age). Seroconversion will be defined as a titer 4-fold higher than the expected fall in maternally derived antibodies, assuming a half-life of 28 days. The initial antibody titer at 6 weeks of age will be used as the starting point for the expected decline in maternal antibody.

This study will compare the immunogenicity of:

1. Sequential dose of intra-dermal f-IPV and bOPV to bOPV alone administered at 6, 10 and 14 weeks of age
2. tOPV to bOPV administered at 6,10 and 14 weeks of age
3. IM IPV to ID f-IPV administered at 6 and 14 weeks of age The answer to these questions will guide the global polio eradication program in designing new routine immunization schedule for children that eliminates the risks of paralysis due to vaccine derived poliovirus (VDPV) from type 2 vaccine poliovirus.

DETAILED DESCRIPTION:
Global polio eradication initiative (GPEI)

In 1988, the World Health Assembly adopted the resolution of polio eradication by 2000. This launched the Global Polio Eradication Initiative (GPEI), spearheaded by World Health Organization (WHO), Rotary International, US Centers for Disease Control and Prevention (CDC) and United Nations Children's Emergency Fund (UNICEF). The major strategies to achieve polio eradication included: 1) provision of 3-4 doses of tOPV to young infants through routine immunization programs; 2) provision of additional doses to all children < 5 years of age through immunization campaigns (supplementary immunization activities or SIAs); 3) surveillance for all cases of acute flaccid paralysis in children <15 years of age; and 4) mop-up immunizations campaigns following the detection of poliovirus circulation.

OPV was the vaccine of choice for polio eradication due to its low cost, ease of administration, ability to induce intestinal immunity and community spread to aid in induction of immunity.

Limitations of trivalent oral polio vaccine (tOPV)

tOPV is a mixture of all three types of polioviruses and there is interference among the strains during intestinal replication. Type 2 especially interferes with uptake of types 1 and 3. tOPV has higher seroconversion rates in industrialized countries compared to that in developing countries. A study conducted in Brazil and Gambia reported tOPV seroconversion rates of 85% for Type 1, 94% for type 2 and 68% for Type 3 with three doses of tOPV. Compared to monovalent OPVs, trivalent OPV has lower seroconversion rates. To address concerns of lower efficacy of tOPV for type 1 and type 3 compared to monovalent vaccines, monovalent vaccines were re-introduced in the polio eradication initiative. Monovalent OPVs are more immunogenic than tOPV. In India, compared to two doses of tOPV given at birth and after 30 days, type-specific seroconversion was significantly higher with two doses of mOPV1 (90% vs. 63%) and mOPV3 (84% vs. 52%). In South Africa, compared to one dose of tOPV given at birth, type-specific seroconversion was significantly higher with one dose of mOPV1 (73% vs. 39%) and mOPV3 (58% vs. 21%).

While the higher immunogenicity of monovalent vaccines compared to trivalent vaccine is highly desirable especially in the presence of a poliovirus outbreak caused by one antigenic type, the monovalent vaccines increase the complication in vaccine selection. Wild type 2 poliovirus was eradicated in 1999 and at the present time there is global circulation of wild poliovirus Type 1 and 3. Weak routine immunization with poor immunization coverage will lead to immunity gaps against all three types of polioviruses. In the presence of Type 1 poliovirus outbreak in a country with weak routine immunization, use of a monovalent Type 1 poliovirus vaccine will contribute to reducing the immunity gap to Type 1 poliovirus, however, this would not address the existing immunity gap to Type 3 poliovirus and vice versa. Additionally, in the presence of an outbreak of Type 1 and Type 3 polioviruses, vaccine selection becomes further complicated. To address these concerns, bivalent OPV (bOPV), mixture of type 1 and type 3, was introduced in the polio eradication program in 2010. The only published clinical trial on bOPV reported that two doses of bOPV given at birth and 30 days later was comparable in immunogenicity to two doses of mOPV1 and mOPV3 and significantly better than two doses of tOPV.

Oral poliovirus vaccines are live attenuated viral vaccines and the vaccine virus in OPV can mutate and acquire neurovirulence causing paralysis either due to vaccine-associated paralytic polio (VAPP) or due to circulating vaccine-derived polioviruses (cVDPV), in which the attenuated vaccine virus not only acquires the ability to cause paralysis but can also circulate similar to wild poliovirus (WPV). The potential of vaccine virus to acquire neurovirulence and cause paralytic poliomyelitis is incompatible with eradication of polio. Therefore, polio eradication will require eventual cessation of all OPVs.

The last case of type 2 WPV (WPV2) was reported in 1999 in India. Type 2 vaccine virus in tOPV is most likely to cause cVDPVs and over 80% of cVDPVs over the past decade have been cVDPV2. Of the estimated 250-500 annual VAPP cases almost 40% are due to type 2. Thus, with the eradication of WPV2 it is imperative to prioritize removal of type 2 containing OPV.

Role of bivalent oral polio vaccine (bOPV) and inactivated polio vaccine (IPV)

The licensing and availability of bivalent OPV (bOPV) containing type 1 and 3 offers the option of an OPV that does not contain OPV2. No studies have assessed the immunogenicity of bOPV when administered in the Expanded Program on Immunization (EPI) schedule of 6, 10 and 14 weeks of age. Additionally, no studies have compared the immunogenicity of bOPV to that of tOPV when administered at 6, 10 and 14 weeks of age. Thus, this comparison has been proposed in this study with inclusion of a bOPV and a tOPV arm.

At the same time, while a switch in routine immunization from tOPV to bOPV has been proposed, there are significant challenges that need to be addressed prior to implementing this possible switch. Removing type 2 OPV from routine immunization will rapidly increase the proportion of population susceptible to type 2. This is turn could facilitate the transmission of cVDPV2 from countries experiencing an outbreak of cVDPV2. Ideally, all cVDPV2 outbreaks will need to be stopped prior to replacement of tOPV with bOPV. Equally important is the need for synchronization of cessation of type 2 OPV globally or regionally to reduce the risk of cVDPV2 importation from countries that continue to use tOPV. The IPV working group of Strategic Advisory Group of Experts on Immunization (SAGE) has endorsed a set of necessary pre-requisites for type 2 OPV cessation and these include: formal validation of absence of WPV2, interruption of cVDPV2 prior to OPV2 cessation, laboratory containment of WPV2, availability of sufficient bOPV for the switch and stockpile of monovalent oral vaccines (mOPV) for outbreak response. At the same time, there is a clear recognition that it would take few more years to achieve the necessary pre-requisites while the balance has already shifted from benefit to risk for type 2 OPV.

Another potential option is to switch from tOPV to IPV but IPV is substantially more expensive than OPV and is not as immunogenic as OPV in inducing mucosal immunity. Hence, the polio eradication program is exploring ways to make IPV affordable for polio eradication that include reducing the number of IPV doses, reducing the antigen content for each dose, manufacturing IPV in developing countries and optimizing other production processes. One of the possible methods of reducing the antigen content of each dose of IPV is to use a fractional injection of IPV (f-IPV) of one-fifth of standard IPV dose given intra-dermally. Compared to intra-muscular injection of IPV, it appears that f-IPV has sub-optimal immunogenicity when administered at 6, 10 and 14 weeks of age (EPI schedule) [ID f-IPV vs IM IPV: Type 1: 53% vs 89%; Type 2: 85% vs 96%; Type 3: 69% vs 99%] though the immunogenicity is comparable when administered at 2, 4 and 6 months of age [ID f-IPV vs IM IPV: Type 1: 97% vs 100%; Type 2: 96% vs 100%; Type 3: 98% vs 100%]. Prior studies have reported that the interval between multiple doses of IPV plays an important role in the immunogenicity of IPV 11. A study conducted in Cuba reported seroconversion rates of 94%, 83% and 100% for Type 1, 2 and 3 respectively with 3 doses of IM IPV administered at 6, 10 and 14 weeks of age. These seroconversion rates were similar to seroconversion observed after 2 doses of IPV administered at 8 and 16 weeks of age (Type 1: 90%; Type 2: 89%; Type 3: 90%). Hence, it is hypothesized that the 1-month interval between the 3 doses in EPI schedule is a major contributor in the sub-optimal immunogenicity of f-IPV compared to the immunogenicity reported with the 2, 4 and 6 month schedule, which has a 2-month interval between doses. As a result in this study the immunogenicity of IM IPV and ID f-IPV administered at 6 and 14 weeks is being assessed where the interval between doses is 2 months.

Justification for this study

There are significant risks associated with switching from tOPV to bOPV in routine immunization. IM IPV is substantially more expensive than tOPV and not as immunogenic in inducing mucosal immunity. These are the principal reasons that prevent use of IM IPV in EPI schedule. ID f-IPV has sub-optimal immunogenicity when used in EPI schedule. Therefore, the polio program needs to test the immunogenicity of combination of poliovirus vaccines as this could potentially address concerns of risks of using bOPV alone and suboptimal immunogenicity of ID f-IPV. Prior studies have shown that IPV and OPV given together as a combination or sequentially with OPV followed by IPV achieves a higher seroconversion than IPV or OPV alone and the mucosal immunity induced by combined IPV and OPV is similar to that induced by OPV. However, seroconversion of sequential f-IPV and bOPV has not yet been determined. Consequently, this study will assess the immunogenicity of a sequential dose of f-IPV and bOPV. Combining bOPV and f-IPV in an immunization schedule has multiple advantages. Firstly, f-IPV will aid in development of Type 2 immunity. Secondly, bOPV combined with f-IPV is likely to be more immunogenic than f-IPV alone. Finally, bOPV is likely to contribute substantially to development of Type 1 and 3 mucosal immunity.

Rationale for the location of the study and the study population

Polio immunization in Bangladesh is provided through the Expanded Program on Immunization to achieve high routine coverage with 3 doses of tOPV in infants younger than 12 months and through National Immunization Days that are usually conducted twice a year. The 3 doses of tOPV through routine immunization services is administered to infants at 6, 10 and 14 weeks of age and WHO/UNICEF estimate coverage of 95% for 2010 with three doses of polio vaccine. With these strategies, Bangladesh interrupted endemic transmission in 2000 and has successfully prevented outbreaks or re-establishment of circulation following importations from neighboring India. With the interruption of polio transmission, Bangladesh is at a critical juncture where it needs to consider steps to reduce the risks associated with emergence of VDPV2. Therefore, it is advantageous to test a potential new combination of existing polio vaccines to reduce risks of VDPV2 emergence in Bangladesh. The results of the study will be applicable in Bangladesh as well as important for the global polio eradication program. ICDDR, B has long-standing expertise in conducting clinical trials and has conducted a polio clinical trial in the proposed site Mirpur, Dhaka. This study reported a seroconversion of 86% for Type1, 97% for Type 2 and 75% for Type 3 after 3 doses of tOPV at 6, 10 and 14 weeks of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants 6-7 weeks of age
* Family that consents for participation in the full length of the study
* Family that is able to understand and comply with planned study procedures

Exclusion Criteria:

* Family that is unable to participate in the full length of the study
* A diagnosis or suspicion of immunodeficiency disorder either in the infant or in an immediate family member
* A diagnosis or suspicion of bleeding disorder that would contraindicate parenteral administration of IPV or collection of blood by venipuncture
* Acute diarrhea, infection or illness at the time of enrollment (6-7 weeks of age) that would require infant's admission to a hospital or would contraindicate provision of OPV per country guidelines
* Acute vomiting and intolerance to liquids within 24 hours before the enrollment visit (6 weeks of age)
* Receipt of any polio vaccine (OPV or IPV) before enrollment based upon documentation or parental recall
* Known allergy/sensitivity or reaction to polio vaccine or contents of polio vaccine
* Infants from multiple births. Infants from multiple are excluded to reduce the potential for contact transmission of vaccine poliovirus. The infant from a multiple birth who is not enrolled is likely to receive routine immunization and transmit vaccine poliovirus to the enrolled infant
* Infants from premature births (<37 weeks of gestation)

Ages: 6 Weeks to 7 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1206 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Seroconversion | Change in antibody titers at 18 weeks of age compared to 6 weeks of age
  The primary analytical approach will be intention-to-treat analysis on enrolled participants who have serological results available on blood specimens collected at 18 weeks of age.
  Reciprocal antibody titers of at least 1:8, the lowest detectable titer, is considered to indicate seropositivity with regards to the presence of poliovirus neutralizing antibodies. Seroconversion is defined as either seronegative participants (<1:8 titers) who become seropositive (≥1:8) or participants who demonstrate a 4-fold change in titers between two specimens, e.g. a change from 1:8 to 1:32. To compare the immunogenicity across study arms, the investigators will compare the proportion of participants who seroconvert by 18 weeks of age. Chi-square tests will be used to test the statistical significance among seroconversion rates across study arms.

SECONDARY OUTCOMES:
Poliovirus shedding in stool | At 19 weeks of age
  Stool specimens collected a week after a challenge dose of tOPV will be analyzed to determine poliovirus shedding. By study arm the investigators will compare proportion of participants shedding poliovirus overall and by type of poliovirus. The investigators will also evaluate quantitative viral shedding (viral titers) and compare these results by study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Abhijeet Anand, MBBS, MPH, Principal Investigator — Centers for Disease Control and Prevention; K. Zaman, MBBS, PhD, Principal Investigator — International Center for Diarrheal Disease Research, Bangladesh
Locations (1):
- Mirpur Health Clinic, Dhaka, Bangladesh